CLINICAL TRIAL: NCT07105670
Title: The Effects of Replacing Red Meat With Alternative Protein Sources on Gut-Derived Metabolites in People With Chronic Kidney Disease
Brief Title: Effects of Replacing High Protein Foods in People With Chronic Kidney Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Sharon Moe, Professor of Medicine, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 25168; K12TR004415 (NIH)
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease Stage 3
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lacto-ovo vegetarian diet (Active Comparator): A lacto-ovo vegetarian diet providing 0.8 g/kg/day of protein.
  Interventions: Other: Controlled dietary intervention
- Red meat diet (Experimental): The lacto-ovo vegetarian diet with 20% of the protein replaced by red meat.
  Interventions: Other: Controlled dietary intervention

INTERVENTIONS:
Other: Controlled dietary intervention — Participants will complete a 2-week baseline period consuming their standard diet without any food or beverages provided followed by a randomized, crossover-controlled feeding study of a lacto-ovo vegetarian diet versus the same diet with 20% of the protein replaced by red meat. In between the two diets, there will be a five-week washout where participants will consume their standard diet without any food or beverages provided.

SUMMARY:
The goal of this crossover clinical trial is to explore the effects of red meat intake on serum and fractional urinary excretion of uremic toxins including trimethylamine N-oxide in people with chronic kidney disease.

DETAILED DESCRIPTION:
This study will be a single-blind crossover, human-feeding study comparing 3 weeks of a lacto-ovo vegetarian diet to the same diet with 20% of the protein replaced by red meat. There will be a 2-week baseline period and a 5-week washout period where participants will consume their typical, self-selected diet. Once eligible, the participant will be randomized to a diet order. The investigators will recruit up to 15 participants. Descriptive statistics (means and standard deviations) will be used to summarize the characteristics of the study population. In general, data will be analyzed using linear mixed-effect models to account for the potential correlation among measurements from the same participant. A power analysis of this pilot study will be conducted based on the estimated interparticipant and intraparticipant variabilities to estimate the required number of participants to detect a certain size of difference with a certain power for a full study.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Male or postmenopausal female
* Stage 3 CKD (eGFR between 30-59ml/min/1.73m^2 by the CKD-EPI equation (without race correction)).
* If eGFR is greater than or equal to 45ml/min/1.73m^2 then albuminuria must be greater than 300mg/g creatinine by spot urine.
* Willing to consume controlled diet for duration of the study
* Willing to collect fecal samples at home

Exclusion Criteria:

* Hemoglobin A1c greater than 7% within previous six months
* Treatment with metformin or insulin within previous three months
* Blood pressure greater than 150/100 mmHg from chart of home on at least two occasions in prior month (can be inclusive of screening visit)
* Change in cardiovascular and/or hypertension medication in the last 30 days
* History of major gastrointestinal disease (e.g. inflammatory bowel disease, uncontrolled irritable bowel syndrome, C. difficile chronic infection, celiac disease, diverticulitis, stomach or duodenal ulcers)
* Known HIV disease
* Hospitalization in the last two months
* Significant recent unintentional weight loss (5% of weight over past three months)
* Cancer or received cancer treatment in the last year (except basal cell carcinoma)
* Prior bariatric surgery (i.e. gastric bypass, sleeve gastrectomy) or restrictive bariatric surgery (i.e. adjustable gastric band)
* Treatment with immunosuppressive medications in the past six months or more than one week of treatment with prednisone greater than 10mg per day in the past three months (or equivalent steroid dose of non-prednisone steroids)
* Recent antibiotic use defined as a single course of antibiotics within the past three months or two or more courses within the past six months
* Known food allergy that would influence the ability to consume the study diets
* History of hyperkalemia defined as greater than 5.5mmol/L on at least two occasions
* Other medical conditions or concerns at the discretion of the investigators

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum trimethylamine N-oxide | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Intra- and interparticipant variability of serum concentrations as measured by high performance liquid chromatography-mass spectrometry

SECONDARY OUTCOMES:
Additional serum uremic toxins | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Including p-cresyl sulfate and indoxyl sulfate measured by high performance liquid chromatography-mass spectrometry
Urinary excretion of uremic toxins | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Measured by a ratio of serum and urine values
Gut microbiota | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Diversity and composition of the gut microbiome
Gastrointestinal symptoms | 13 Weeks (collections in week 2, 5, 10, and 13 which corresponds to before and during the last week of each of the three-week controlled diet periods).
  Measured at the end of each study period by the Gastrointestinal Symptom Rating Scale. This is a 15-item questionnaire that includes five domains. Each item is scored from 1 to 7 and the mean score in each domain is presented.
Stool consistency | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Measured on a scale from 1 to 7 using the Bristol Stool Scale/Chart.
Blood pressure | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Arterial Stiffness | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Carotid-femoral pulse wave velocity
Height | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Weight | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Handgrip Strength | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Total cholesterol | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
High density lipoprotein | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Low Density Lipoprotein | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Triglycerides | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Apolipoprotein B | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Blood glucose | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
  Fasting blood glucose
Serum calcium | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Serum Potassium | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Serum bicarbonate | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Subjective global assessment | 13 Weeks (collections in week 2, 5, 10, 13 which corresponds to before and during the last week of each of the three-week controlled diet periods).
  Scored on a scale from 1-7 (severely malnourished to well nourished)
Albumin to creatinine ratio | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Blood urea nitrogen | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Creatinine | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Serum Phosphate | 13 Weeks (collections in week 1, 2, 4, 5, 9, 10, 12, 13 which corresponds to before and during the last two weeks of each of the three-week controlled diet periods).
Urinary phosphorus excretion | 13 Weeks (collections in week 2, 5, 10, 13 which corresponds to before and after each of the three-week controlled diet periods).
  From 24-hour urine collection

CONTACTS AND LOCATIONS:
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No